CLINICAL TRIAL: NCT04572542
Title: Camrelizumab Combined With Apatinib Mesylate Tablets and Nab-paclitaxel in the Second-line Treatment of Advanced Gastric Cancer： a Single-arm, Multicenter， Prospective Phase II Study
Brief Title: Camrelizumab Combined With Apatinib Mesylate Tablets and Nab-paclitaxel in the Second-line Treatment of Advanced Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Arise-FJ-G202
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Locally Advanced or Metastatic Gastric Adenocarcinoma
MeSH Terms: interventions — camrelizumab; apatinib; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab + Apatinib + nab-paclitaxel (Experimental): Camrelizumab combined with Apatinib mesylate tablets and nab-paclitaxel in the second-line treatment of advanced gastric cancer
  Interventions: Drug: Camrelizumab; Drug: Apatinib Mesylate; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab One course will last 21 days.Given once every 3 weeks at a dose of 200 mg
Drug: Apatinib Mesylate — Apatinib One course will last 21 days.Oral administration at a dose of 250 mg everyday
Drug: nab-paclitaxel — nab-paclitaxel One course will last 21 days。Given twice every 3 weeks at a dose of 125 mg/m2

SUMMARY:
To evaluate the clinical efficacy and safety of camrelizumab combined with apatinib mesylate and nab-paclitaxel .

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years of age
* Gastric adenocarcinoma (papillary adenocarcinoma pap, tubular adenocarcinoma tub, mucinous adenocarcinoma muc, sig-ring cell carcinoma sig, poorly differentiated adenocarcinoma por) confirmed by pathology (including histology or cytology) is an unresectable locally advanced or metastatic (stage IV) tumor.
* For patients with advanced gastric cancer who had received standard first-line treatment in the past, the interval of the last chemotherapy should be more than 1 month .
* Measurable lesions at least should be detected by CT/MRI examination in accordance with the RECIST1.1.（CT scan of tumor lesion length≥10mm，CT scan short diameter≥15mm，scan slice thicknes 5mm）.
* ECOG（Eastern Cooperative Oncology Group）:0-2 scores.
* The expected survival time is more than 3 months.
* The damage caused by subjects receiving other treatments has recovered, including receiving nitroso or mitomycin at intervals >=6 weeks; Received other cytotoxic drugs, radiotherapy or surgery >=4 weeks, and the wound had completely healed .
* Patients with adequate organ function at the time of enrollment as defined below:

  1. Blood routine examination standard (without blood transfusion within 14 days before enrollment):

     1. HB >=90g/L;
     2. WBC >=3.5x10^9/L;
     3. ANC >=1.5x10^9/L;
     4. PLT >=75x10^9/L;
  2. Biochemical examination shall meet the following standards: a.BIL <1.25 ULN; b.ALT and AST< 2.5 ULN; If liver metastasis is present ALT and AST< 5 ULN; c.Serum creatinine Cr <=1 ULN; Serum creatinine >50ml/min (Cockcroft-Gault math);
* Women of childbearing age must have a pregnancy test in 7 days before entering the group (in serum), and the results were negative, and willing to use appropriate contraception during the study period and the last 8 weeks after giving drug test; men should have the surgical sterilization, or adopt the appropriate contraceptive methods during the test and the last 8 weeks after giving drug test.
* Participants is willing to participate in this study, sign the informed consent, have good compliance, cooperate with follow-up.

Exclusion Criteria:

* Patients with chemotherapy and contraindications to Apatinib mesylate.
* Previous history of receiving purpuranoidins, Apatinib mesylate or other antiangiogenic drugs, Camrelizumab or other immunotherapy.
* Pregnant or lactating women.
* Those who participated in other clinical studies and did not recover from toxic reactions within 1 month before enrollment.
* Except for other malignant tumors, basal cell carcinoma of the skin and cervical cancer in situ in the past 5 years.
* Accompanied by serious heart, lung, liver, kidney disease; Have nerve, mental disease; Jaundice or obstruction of the digestive tract with severe infection
* The presence of uncontrolled or symptomatic active central nervous system (CNS) metastases may manifest as the presence of clinical symptoms, cerebral edema, spinal cord compression meningitis, ptosis, and/or progressive growth. After adequate treatment for CNS metastases, neurological symptoms can return to baseline at least 2 weeks prior to randomization (residual signs or symptoms associated with CNS treatment can be enrolled in the study. In addition, subjects must either discontinue corticosteroids or receive prednisone (or an equivalent dose of other corticosteroids) at a steady dose of ≤ 10 mg/d or a gradually reduced dose for at least 2 weeks prior to randomization.
* The blood pressure of patients with hypertension cannot be reduced to the normal range by the antihypertensive drugs (systolic pressure >140 mmHg, diastolic pressure >90 mmHg)
* With Ⅰ magnitude of coronary heart disease, arrhythmia (including QTc protracted between male > 450 ms, women > 470 ms) and cardiac insufficiency
* Patients have a clear tendency with gastrointestinal bleeding, including the following situation: local active ulcerative lesions, and fecal occult blood (+ +); with melena and hematemesis history in 2 months; and patients with fecal occult blood (+) and unresected gastric primary tumor; patients with the risk of bleeding should take the gastroscopy test, if it is the gastric cancer, and researchers believe that may results in massive digestive tract hemorrhage；coagulation dysfunction (INR(international normalized ratio)>1.5, APTT(activated partial thromboplastin time)>1.5 ULN), with bleeding tendency;
* Patients with a history of cardiovascular and cerebrovascular diseases who are still taking oral thrombolytic drugs or anticoagulant drugs
* Patients are positive of urine protein (urine protein detection 2+ or above, or 24 hours urine protein quantitative >1.0g).
* Presence of any active, known or suspected autoimmune disease. Allowed to be included in a stable state, do not need systemic immunosuppression treatment of subjects: such as Ⅰ diabetes, only need to hormone replacement therapy for hypothyroidism and without systemic treatment of skin disease (for example, vitiligo, psoriasis, and hair loss).
* A history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency disorders, or a history of organ transplantation and allogeneic bone marrow transplantation.
* Patients with other concomitant diseases that, at the investigator's discretion, pose a serious risk to patient safety or affect patient completion of the study.
* Patients with uncontrolled epilepsy, central nervous system disease, or mental disorders whose clinical severity, as determined by the investigator, may prevent the signing of the informed consent or have multiple factors that affect oral medications (such as inability to swallow, persistent uncontrolled nausea and vomiting, chronic diarrhea, and intestinal obstruction).
* A person who has previously been allergic to any component of Camrelizumab or to any component of the drug under study.
* The researchers consider those who were not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | one year
  Objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumours (RECIST) version. 1.1, and immune-related (ir) RECIST

SECONDARY OUTCOMES:
Disease Control Rate（DCR） | one year
  Disease Control Rate（DCR） according to Response Evaluation Criteria in Solid Tumours (RECIST) version. 1.1, and immune-related (ir) RECIST

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China